CLINICAL TRIAL: NCT00006526
Title: Coronary Calcification Progression Study
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 951; R01HL063264 (NIH)
Record Dates: First submitted 2000-11-28; First posted 2000-11-28 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases

SUMMARY:
To investigate use of Fast Gated Helical Computed Tomography (FGHCT) measures of coronary artery calcium (CAC), FGHCT-CAC, for discrimination of coronary artery disease (CAD) and to quantify progression of coronary artery calcium over time.

DETAILED DESCRIPTION:
BACKGROUND:

While advances have been made in control of some coronary heart disease (CHD) risk factors, especially smoking and high dietary fat intake, much of the decline in age-adjusted CHD mortality rates has been due to medical treatment and procedural interventions for overt CHD as well as hypertension and hypercholesterolemia. In this context, the availability of an inexpensive, sensitive and specific method for noninvasive detection of both early coronary atherosclerosis and asymptomatic but advanced CHD could allow beneficial treatments to be targeted at many high-risk individuals. The study was designed to determine whether fast-gated helical computed tomography (FGHCT), a more advanced and readily-available variant of a technique (EBCT) that has not achieved its full promise, could play such a role.

DESIGN NARRATIVE:

Dr. Crouse and his colleagues augmented ongoing case-control studies, HL35333, "Carotid Atherosclerosis Progression Study" and HL59503, "Vascular Disease, Structure and Function". HL35333 comprises 280 symptomatic individuals > 45 years equally divided between men and women, half with and half without angiographically defined coronary artery disease evaluated for risk factors and extracranial carotid intimal-medial thickness (ECIMT, with B-mode ultrasound) at baseline and yearly for three years. The grant has quantified the associations of coronary artery disease and coronary artery disease risk factors for ECIMT and its progression. HL59503 quantifies flow-mediated brachial artery reactivity (FM-BAR) in this cohort. Literature review suggests that while ECIMT predicts coronary artery disease status in clinical samples it does less well in asymptomatic samples; longitudinal data (CLAS study) suggest that progression of ECIMT best predicted incident coronary artery disease, and Electron Beam Computed Tomography (EBCT) quantification of Coronary Artery Calcium (CAC) likely has even greater discriminatory power for coronary artery disease than ECIMT. However, EBCT has limited accessibility.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-07; Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Crouse — Wake Forest University